CLINICAL TRIAL: NCT02115568
Title: A Registry to Assess the Ongoing Safety for Subjects That Have Been Randomized and Completed a Juventas Sponsored Heart Failure Protocol Under IND # 14203
Brief Title: Registry to Assess Safety for Subjects That Have Completed a Juventas Sponsored HF Protocol Under IND # 14203
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Juventas Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: JTCS-005
Record Dates: First submitted 2014-04-07; First posted 2014-04-16 (Estimated); Last update posted 2014-04-16 (Estimated); Status verified 2014-04

CONDITIONS: Ischemic Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Long-term safety follow-up: To be eligible, subjects must have actively participated in a Juventas (JVS-100) sponsored trial under IND 14203.

SUMMARY:
This is an exploratory registry that will include subjects who have been randomized to receive JVS-100 treatment (at one of multiple doses) or placebo by one of a number of delivery systems (e.g. endomyocardial injection, retrograde infusion) in a previous Juventas clinical trial.

DETAILED DESCRIPTION:
This Registry will assess the ongoing safety of subjects including morbidity/mortality parameters as they relate to heart failure and track any newly diagnosed malignancies. The logistics of the study are as follows: to be eligible, subjects must have actively participated in a Juventas sponsored trial under IND 14203. After consent, subjects will be followed for up to three years post receipt of investigational product during which time they will receive phone calls (every 3 months) from the study site asking about their health. Questions will be aimed at cardiovascular related events including:

* Hospitalizations
* ER Visits
* Unscheduled visits with Cardiologist
* Newly diagnosed malignancies Serious Adverse Events (SAEs) will not be reported in this study; however, data pertaining to such events will be captured (i.e. date of admission and diagnosis.). Data will be captured on paper CRFs, collected by Juventas (or their designee) and will be entered into a clinical database for analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participated in and completed a Juventas sponsored heart failure study under IND 14203

Exclusion Criteria:

* Unwillingness to sign informed consent form
* Unwillingness or inability to receive phone calls for required follow up assessments
* Subjects actively participating in another regenerative medicine trial should be discussed with sponsor prior to enrollment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population eligible for the proposed Registry will be subjects who have completed a Juventas sponsored heart failure study under IND 14203. The patient population will primarily be comprised of symptomatic systolic heart failure patients due to ischemic etiology.
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2014-01; Primary Completion 2017-01 (Estimated); Study Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Morbidity/Mortality | 3 years
  A questionnaire will be used to assess the ongoing safety of subjects including morbidity/mortality parameters as they relate to heart failure.

SECONDARY OUTCOMES:
Newly diagnosed malignancies | 3 years
  A questionnaire will be used to track any newly diagnosed malignancies.

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Cardiology, P.C., Birmingham, Alabama
  - University of Florida, Gainsville, Florida
  - Pepin Heart Institute, Tampa, Florida
  - Iowa Heart Center, Des Moines, Iowa
  - University of Kentucky Gill Heart Institute, Lexington, Kentucky
  - Johns Hopkins University, Baltimore, Maryland
  - Michigan Cardiovascular Institute, Saginaw, Michigan
  - Saint Luke's Hospital of Kansas City, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - Columbia University Medical Center, New York, New York
  - Summa Health System, Akron, Ohio
  - The Carl and Edyth Lindner Center for Research & Education at The Christ Hospital, Cincinnati, Ohio
  - University of Pennsylvania Health System, Philadelphia, Pennsylvania
  - University of Utah, Salt Lake City, Utah